CLINICAL TRIAL: NCT03472235
Title: Combined Trichlotoaceticacid and Microneedle Versus Trichlroacetic Acid Alone in the Treatment of Melasma
Brief Title: Microneedle and Trichloroaceticacid in Treatment of Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Hamed, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTTM
Record Dates: First submitted 2018-02-07; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-02

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: TCA peeling session: Facial skin will be cleansed with tap water and degreased by rubbing with an alcohol sponge .
  Then TCA 25% will be applied to the whole face by cotton tipped applicator or gauze pad. The entire face will be treated until complete frosting occur.
  The patients will be instructed to wash their faces to decrease the burning sensation.
  Combined session: starts with microneedling using microneedling device (Dermapen) The skin of each patient is cleaned with anti septic solution and anesthetic cream may be applied to lessen discomfort.
  (Dermapen) will be applied on the lesional skin in four direction, vertical, horizontal and in the two diagonal until pin point bleeding occur which will be gently massaged .
  After 10 minutes TCA peeling will be applied TCA peeling will be done for 8 session with 2 weeks interval between each session.
  Microneedling will be done for 4session with 4 weeks interval between each session.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): include 20 patients will be treated with TCA25% +microneedle 8 sessions for TCA 25 peel and 4 sessions for microneedle (derma pen).
  Interventions: Device: Microneedle
- B (Active Comparator): include 20 patient will be treated with TCA 25% only ( 8 sessions)
  Interventions: Device: Microneedle

INTERVENTIONS:
Device: Microneedle — TCA peeling session: Facial skin will be cleansed with tap water and degreased by rubbing with an alcohol sponge .
  Then TCA 25% will be applied to the whole face by cotton tipped applicator or gauze pad. The entire face will be treated until complete frosting occur.
  The patients will be instructed to wash their faces to decrease the burning sensation.
  Combined session: starts with microneedle using microneedle device (Derma pen) The skin of each patient is cleaned with anti septic solution and anesthetic cream may be applied to lessen discomfort.
  (Dermapen) will be applied on the lesional skin in four direction, vertical, horizontal and in the two diagonal until pin point bleeding occur which will be gently massaged .
  After 10 minutes TCA peeling will be applied TCA peeling will be done for 8 session with 2 weeks interval between each session.
  Microneedle will be done for 4session with 4 weeks interval between each session.

SUMMARY:
Melasma is an acquired disorder of hyperpigmentation characterised by blotchy, light-to-dark brown macules distributed symmetrically on the sun-exposed parts of the body.

Although many factors have been proposed to have a role in pathogenesis, the exact ethology is yet to be understood. The most commonly identifiable risk factors include ultraviolet radiation, genetic predisposition, pregnancy, oral contraceptives, thyroid disease and drugs like antiepileptic. The excessive pigmentation has been attributed to both melanocytosis (increased number of melanocytes) as well as melano genesis (excess production of melanin) as confirmed in a histopathological study on Asian patients.] Furthermore, a vascular component has also been proposed to play a role in the pathogenesis of melisma. Kim et al. have found that lesion melasma skin had greater expression of the vascular endothelial growth factor in keratinocytes compared to nearby nonlesional skin.

DETAILED DESCRIPTION:
As regards management, the therapeutic options range from photoprotection, topical hypopigmenting agents, chemical peels and lasers. There are variety of less-tried systemic agents like fish oil, green tea and . Although no single agent has proved to be effective for all patients, a combination of two or three agents is often tried to achieve optimum results.

Chemical peeling is the application of a chemical agent to the skin, which causes the controlled destruction of a part or of the entire epidermis, with or without the dermis, leading to exfoliation and removal of superficial lesions, followed by the regeneration of new epidermal and dermal tissues.

Chemical peels are a well-known modality of treatment for melasma. The basic mechanism of the action of chemical peels in melasma is the removal of unwanted melanin by causing a controlled chemical burn to the skin.

Trichlroacetic acid peeling has been the gold standard in chemical peeling for many decades.

For superficial peels Trichlroacetic acid 10% to 25% are used. some authors consider up to 35% Trichlroacetic acid as also a superficial.

Skin microneedling is a technique predominantly used to improve the appearance of cutaneous scarring and photo damage.

Fine needles puncture the skin, resulting in increased dermal elastin and collagen, collagen remodelling, and thickening of the epidermis and dermis. Additionally, skin needling creates small channels, which increase the absorption of topically applied preparations A property which has been used in various dermatological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Both sex will be included Age range from 18- 50 yrs.' old Patients with realistic expectations.

Exclusion Criteria:

* patients taking oral contraceptive pills. patients with history of polycystic ovary. pregnant and lactating females. patients with active infection. patients on isotretinoin. patients with history of keloids,or hypertrophic scars.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-05 (Estimated); Primary Completion 2019-04-05 (Estimated); Study Completion 2020-04-05 (Estimated)

PRIMARY OUTCOMES:
Scoring of the patients according to modified melasma are abd severity index [mMASI] Scoring before and After last session will be done by 1 month | 1 month after last session
  Efficacy of the treatment =(mMASIscorebefor -mMASIscoreafter)/mMASIscore before x100.
  Clinical efficacy was categorized into :
  Excellent response: if morethan 75%fall in [mMASI] score. Very good response:if 50-75%fall in ]mMASI[score . Good respone: if 25-50%fall in ]mMASI[score. Poor response: if less25%fall in mMASIscore. No response: when there was no change in [mMASI] score at the end of the therapy.
  Efficacy of the treatment =(mMASIscorebefor -mMASIscoreafter)/mMASIscore before x100.
  Clinical efficacy was categorized into :
  Excellent response: if morethan 75%fall in [mMASI] score. Very goodresponse:if 50-75%fall in ]mMASI[score . Good respone: if 25-50%fall in ]mMASI[score. Poor response: if less25%fall in mMASIscore. No response: when there was no change in [mMASI] score at the end of the therapy.
[mMASI] Scoring before and After last session will be done by 3 months | 3 months after last session
  before x100.
  Clinical efficacy was categorized into :
  Excellent response: if morethan 75%fall in [mMASI] score. Very good response:if 50-75%fall in ]mMASI[score . Good respone: if 25-50%fall in ]mMASI[score. Poor response: if less25%fall in mMASIscore. No response: when there was no change in [mMASI] score at the end of the therapy.
  Efficacy of the treatment =(mMASIscorebefor -mMASIscoreafter)/mMASIscore before x100.
  Clinical efficacy was categorized into :
  Excellent response: if morethan 75%fall in [mMASI] score. Very goodresponse:if 50-75%fall in ]mMASI[score . Good respone: if 25-50%fall in ]mMASI[score. Poor response: if less25%fall in mMASIscore. No response: when there was no c

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheth VM, Pandya AG. Melasma: a comprehensive update: part II. J Am Acad Dermatol. 2011 Oct;65(4):699-714. doi: 10.1016/j.jaad.2011.06.001. PMID 21920242